CLINICAL TRIAL: NCT07061028
Title: The Effects of Progressive Muscle Relaxation on Pain Intensity, Pain Catastrophizing, and Quality of Life in Patients With End Stage Renal Disease: A Randomized Controlled Study
Brief Title: Effect of PMR on Pain In Patients With ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate Peofessor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/136
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Progressive Muscle Relaxation; End Stage Kidney Disease; Pain; Pain Catastrophizing; Quality of Life
MeSH Terms: conditions — Kidney Failure, Chronic; Pain | interventions — Autogenic Training; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (Experimental): This group received five weekly 30-minute sessions of Progressive Muscle Relaxation (PMR) based on the ABC relaxation theory. The PMR protocol developed by Smith (2005) involve tense-and-release exercises for 11 different muscle groups, including hands, arms, sides, back, shoulders, face, neck, stomach, chest, legs, and feet. For five to ten seconds, each muscle group is contracted, and for twenty to thirty seconds, it is relaxed. The sensations of stress and relaxation were the participants' main concern. To release any residual tension, they looked at each muscle group after the workout. With the exception of the time needed for measurements and instructions, the entire operation took roughly thirty minutes.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Waitlist Control Group (Other): The control group received no intervention from the researcher during the study. However, following the intervention, the control group participants were given the audio recordings of the intervention protocol along with an explanation of them.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — This intervention involves five weekly 30-minute sessions of Progressive Muscle Relaxation (PMR) based on the ABC relaxation theory. The PMR protocol developed by Smith (2005) involve tense-and-release exercises for 11 different muscle groups, including hands, arms, sides, back, shoulders, face, neck, stomach, chest, legs, and feet. For five to ten seconds, each muscle group is contracted, and for twenty to thirty seconds, it is relaxed. The sensations of stress and relaxation were the participants' main concern. To release any residual tension, they looked at each muscle group after the workout. With the exception of the time needed for measurements and instructions, the entire operation took roughly thirty minutes.
  Arms: Progressive Muscle Relaxation
Other: Control Group — The control group received no intervention from the researcher during the study. However, following the intervention, the control group participants were given the audio recordings of the intervention protocol along with an explanation of them.
  Arms: Waitlist Control Group

SUMMARY:
Background: Patients with chronic end-stage renal disease (ESRD) commonly experience chronic pain, which significantly impair their quality of life. This pain is often exacerbated by maladaptive cognitive appraisals, in particular pain catastrophizing. This study investigated the effectiveness of progressive muscle relaxation (PMR) on pain intensity, pain catastrophizing, and health-related quality of life on patients undergoing with ESRD.

Methods: This randomized controlled parallel study was conducted in a governmental hospital in Jordan in 2024. Participants (N= 104) were randomly assigned to an experimental group offered five sessions of 30 minutes of PMR per week over a total period of five weeks and a control group, which receives standard treatment. The outcomes were measured by Arabic validated scales such as the Pain Catastrophizing Scale, Numerical Pain Rating Scale and the Renal Disease Quality of Life questionnaire at baseline and the end of the intervention.

DETAILED DESCRIPTION:
Patients with chronic end-stage renal disease (ESRD) commonly experience chronic pain, which significantly impair their quality of life. This pain is often exacerbated by maladaptive cognitive appraisals, in particular pain catastrophizing. This study investigated the effectiveness of progressive muscle relaxation (PMR) on pain intensity, pain catastrophizing, and health-related quality of life on patients undergoing with ESRD.

This study using a pretest-post-test randomized controlled parallel design was conducted in a Dialysis facility in a Government Military Hospitals. This facility is the biggest in the middle east that includes 58 dialysis machines and treats 2,200-2,240 patients monthly. The participants were chosen by a convenience sampling method and then randomly allocated into experimental and control groups. Research assistant who did not participate in any phase of the study (e.g. recruitment or measurement) performed the participants' allocation using a cluster random assignment method explained below.

The sample size was calculated using G*power 3.1.9.4. The estimated sample size was 102 given an independent t-test, a medium effect size of 0.5, an alpha of 0.05, and a power of 0.8. Considering a 15% attrition rate, 117 participants are needed for the sample. The final necessary sample size was 120 individuals after 3 persons were added to be more cautious. Out of the 170 individuals that had their eligibility evaluated, 120 were found to be eligible and consented to take part. 104 of them finished the study, and their data was analysed. Due to health concerns, the remaining 16 participants decided to leave the study prior to the collection of baseline data.

After getting the approval of the Institutional Research Board (IRB), the research investigator approached hospital management requesting them to allow the study to be carried out at their hospital. Upon consent, the researcher interviewed the subjects individually on their study objectives and processes. The informed consent statement was forwarded to all the participants who had agreed to participate in the research. The participants were then randomly assigned to the experimental group and the control group using a cluster random assignment to avoid contamination. To implement this assignment approach, a list of participants who met the criteria for the research was made, along with their shifts (A, B, and C). Participants received hemodialysis three times a week on either Sunday, Tuesday, and Thursday (STT) or Monday, Wednesday, and Saturday (MWS). The above arrangement resulted in six clusters: two shifts per week (STT or MWS) × three shifts per day (A, B, and C). The clusters (STT Shift A, 2) STT Shift B, 3) STT Shift C, 4) MWS Shift A, 5) MWS Shift B, and 6) MMWS Shift C were defined by a mixture of hemodialysis days and shifts. Listing all six clusters-each with twenty subjects according to the sample size calculation-was an initial procedure. Following that, these clusters were randomly assigned to the control or experimental groups. Randomizing participants was carried out using a random number generation technique to ensure an unbiased assignment. This random assignment method was used by an investigator who had no involvement in recruiting participants and was blind to the participant list.

After randomization, baseline assessments of the study sociodemographics and dependent variables were conducted in the hemodialysis unit before the intervention started. At the end of the intervention, which occurred five weeks following the actual MBI training, the study dependent variables were assessed again. A qualified research assistant collected the data without taking part in other study components. A qualified research assistant collected the data without taking part in other study components. This research assistant has a strong background in nephrology and is a registered nurse. Every measurement in the hemodialysis unit was conducted in private, with similar settings (e.g., temperature) and conditions (e.g., sitting position). There was nobody there when they finished the questionnaire.

This study employed five weekly 30-minute sessions of Progressive Muscle Relaxation (PMR) based on the ABC relaxation theory. The PMR intervention involve tense-and-release exercises for 11 different muscle groups, including hands, arms, sides, back, shoulders, face, neck, stomach, chest, legs, and feet. For five to ten seconds, each muscle group is contracted, and for twenty to thirty seconds, it is relaxed. The sensations of stress and relaxation were the participants' main concern. To release any residual tension, they looked at each muscle group after the workout. With the exception of the time needed for measurements and instructions, the entire operation took roughly thirty minutes.

Participants in the experimental group attended three weekly PMR sessions during their five weeks of hemodialysis. In order to allow participants to practice the PMR procedure during hemodialysis sessions, it was recorded on audio. These recordings were provided to them via email or WhatsApp, depending on their option. This audio recording was made utilizing Smith's protocol by a certified study researcher who holds a higher degree in nursing and has extensive experience practicing and delivering mind-body therapies. The audio recording was confirmed and authenticated by two psychologists with strong PMR backgrounds. The researcher managed any interruptions, kept the PMR delivery under control, protected confidentiality, and made sure they could practice efficiently. Although it was not required, participants were encouraged to practice the PMR at home during the five-week trial period. Prior to the trial, participants in both groups were told to stick to their regular schedules and refrain from pursuing alternative or psychiatric therapy to elevate their mood. They were also requested to inform the researcher if they decided to seek such treatments during the study time. They were also requested to notify the researcher if they used analgesics during the study period.

Before the intervention started, a face-to-face instructional session was held to help participants better understand it. Consequently, the participants in the experimental group attended an additional 2-hour education session during which the researcher gave them thorough information regarding the purpose and approach of the intervention. During the workshop, participants learnt the basics of the PMR program and were given a detailed walkthrough of the full intervention process. Participants were encouraged to ask questions and take part in conversations to ensure they understood the intervention. The control group received no interaction from the researcher. However, following the conclusion of the investigation, the control group participants were given the audio recordings of the intervention protocol along with an explanation of them.

Version 25 of the statistical package for social science was used to analyze our data. To provide an overview of the study results, descriptive statistics were applied. Because the data was not normally distributed, we described categorical variables with frequency and percentage and continuous variables with median and IQR. Histogram, the Shapiro-Wilk test, and skewness and kurtosis indices were used to examine the normality across groups. The homogeneity of variance was examined using Levene's test. If continuous variables' data did not follow the normal distribution and had unequal variances, non-parametric tests such as Mann-Whitney U tests and Wilcoxon Signed Ranks Test replaced parametric tests including independent tests and dependet t-tests respectively.

A chi-square test was performed to study whether there were baseline differences on sociodemographic categorical variables between the study groups. Mann-Whitney U tests were used to compare the difference between two independent groups at baseline and after the intervention as normality and/or homogeneity of variance were violated. To find out if the mean scores improved within the study groups, a Wilcoxon Signed Ranks Test was run, since not all data followed a normal distribution.

This study obtained a approval by the IRB at Jordan University of Science and Technology. The consenting participants were made to read and sign a consent form after which they were allowed to engage in the study. They were assured that they would not face any impact on their access to care in case they refuse to participate. The participants were informed that their names were converted to numbers because of their anonymity and that the research information would be stored safely in an encrypted file cabinet which can only be accessed by the investigators. No eligible patient was excluded due to her or his racio- ethnic background. The intervention was stopped, and the doctor was notified right away if the participants experienced discomfort.

ELIGIBILITY:
Inclusion Criteria:

* The patients with ESRD who had a smartphone
* aged eighteen years or above
* and received hemodialysis at least thrice a week

Exclusion Criteria:

* The patients with ESRD patients who received psychotherapy
* or took regular psychopharmacological and analgesic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
The Arabic Pain Catastrophizing Scale | From enrollment to the end of treatment at 6 weeks
  The Arabic Pain Catastrophizing Scale (PCS) was used to measure pain catastrophizing in the study. It consists of 13 items that evaluate an individual's thoughts and emotions connected to pain. Three aspects of pain catastrophizing are measured by PCS: helplessness (6 items) magnification (3 items) and rumination (4 items). Patients rate how often they experience the above thoughts and sensations when they are in pain. They use a 5-point Likert-type scale, ranging from 0 (not at all) 1 to 4 (all the time). By adding together, the scores for each question, one may get the subscale scores. These scores are between 0 to 52, with higher scores are indicative of a greater pain catastrophizing. A reliable and valid method for assessing catastrophizing in chronic pain patients who speak Arabic is the Arabic version of the Pain Catastrophizing Scale (PCS). The scale demonstrated strong internal consistency, with a Cronbach's α of 0.94.
Visual Analog Scale (VAS) | From enrollment to the end of intervention at 6 weeks
  The scale asks respondents to select the value (between 0 and 10) which most closely represents their level of pain. High test-retest reliability has been demonstrated by both literate and illiterate rheumatoid arthritis patients (r = 0.96 and 0.95, respectively). With correlation ranging from 0.86 to 0.95, the NPRS was found to have a strong association with the VAS for construct validity among individuals with chronic pain disorders (pain that lasts a minimum of six months). The scale has been found to be a valid and reliable tool for assessing pain severity in Arabic-speaking nations.
Arabic version of the kidney disease-related Quality of Life questionnaire | From enrollment to the end of intervention at 6 weeks
  Quality of life was assessed using the Arabic version of the kidney disease-related Quality of Life questionnaire (KDQOL-36). It comprises four subscales: generic core [Physical Component Summary (PCS, 12 items) and mental component summary (MCS, 12 items); symptoms and issues (12 items); burden of renal disease (4 items); and impacts of kidney disease (8 items) (Elamin et al., 2019). The raw, pre-coded numerical values of each item are linearly transformed into a scale ranging from 0 to 100, where higher numbers denote a higher quality of life. Positive psychometric characteristics were found in Arabic patients with chronic renal insufficiency using the scale's Arabic version. With a Cronbach's alpha of 0.81, the KDQOL-36 translation demonstrated high internal reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology/ King Abdullah University Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith, J. C. (2005). Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. Springer Publishing Company.
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7(4), 524-532. https://doi.org/10.1037/1040-3590.7.4.524
- [Background] Terkawi AS, Sullivan M, Abolkhair A, Al-Zhahrani T, Terkawi RS, Alasfar EM, Khait SSA, Elkabbani A, Kabbani N, Altirkawi KA, Tsang S. Development and validation of Arabic version of the pain catastrophizing scale. Saudi J Anaesth. 2017 May;11(Suppl 1):S63-S70. doi: 10.4103/sja.SJA_130_17. PMID 28616005
- [Background] Zhang C, Zhang Z, Li Y, Feng C, Meng H, Gao Y, Lo WLA, Wang C. Pain Catastrophizing Is Related to Static Postural Control Impairment in Patients with Nonspecific Chronic Low Back Pain: A Cross-Sectional Study. Pain Res Manag. 2020 Oct 28;2020:9629526. doi: 10.1155/2020/9629526. eCollection 2020. PMID 33193926
- [Background] Wolff B, Burns JW, Quartana PJ, Lofland K, Bruehl S, Chung OY. Pain catastrophizing, physiological indexes, and chronic pain severity: tests of mediation and moderation models. J Behav Med. 2008 Apr;31(2):105-14. doi: 10.1007/s10865-007-9138-z. PMID 18158618
- [Background] Kesik G, Ozdemir L, Mungan Ozturk S. The Effects of Relaxation Techniques on Pain, Fatigue, and Kinesiophobia in Multiple Sclerosis Patients: A 3-Arm Randomized Trial. J Neurosci Nurs. 2022 Apr 1;54(2):86-91. doi: 10.1097/JNN.0000000000000620. PMID 35149625
- [Background] Kazak A, Ozkaraman A. The Effect of Progressive Muscle Relaxation Exercises on Pain on Patients with Sickle Cell Disease: Randomized Controlled Study. Pain Manag Nurs. 2021 Apr;22(2):177-183. doi: 10.1016/j.pmn.2020.02.069. Epub 2020 Mar 26. PMID 32224022
- [Background] Karakus A, Uzelpasaci E, Akyurek G. The comparative effectiveness of progressive relaxation training on pain characteristics, attack frequency, activity self-efficacy, and pain-related disability in women with episodic tension-type headache and migraine. PLoS One. 2025 Apr 28;20(4):e0320575. doi: 10.1371/journal.pone.0320575. eCollection 2025. PMID 40293994
- [Background] Kaplan Serin E, Ovayolu N, Ovayolu O. The Effect of Progressive Relaxation Exercises on Pain, Fatigue, and Quality of Life in Dialysis Patients. Holist Nurs Pract. 2020 Mar/Apr;34(2):121-128. doi: 10.1097/HNP.0000000000000347. PMID 31567304
- [Background] Izgu N, Gok Metin Z, Karadas C, Ozdemir L, Metinarikan N, Corapcioglu D. Progressive Muscle Relaxation and Mindfulness Meditation on Neuropathic Pain, Fatigue, and Quality of Life in Patients With Type 2 Diabetes: A Randomized Clinical Trial. J Nurs Scholarsh. 2020 Sep;52(5):476-487. doi: 10.1111/jnu.12580. Epub 2020 Jun 13. PMID 32536026
- [Background] He CC, Lin DM, Liu HZ, Wang FF, Guo XF, Zhang XB, Ai YQ, Meng LM. Nonpharmacological Interventions for Management of the Pain-Fatigue-Sleep Disturbance Symptom Cluster in Breast Cancer Patients: A Systematic Review and Network Meta-Analysis of Randomized Controlled Trials. J Pain Res. 2023 Aug 7;16:2713-2728. doi: 10.2147/JPR.S409798. eCollection 2023. PMID 37577159
- [Background] Fonseca das Neves J, Kornacka M, Serra E, Rollin N, Kosinski T, Marechal V, Jehel L, Rusinek S. The impact of rumination on fibromyalgia pain after physical activity: an experimental study. Sci Rep. 2023 Nov 22;13(1):20523. doi: 10.1038/s41598-023-47414-z. PMID 37993555
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Feldmann M, Hein HJ, Voderholzer U, Doerr R, Hoff T, Langs G, Herzog P, Kaiser T, Rief W, Riecke J, Brakemeier EL. Cognitive Change and Relaxation as Key Mechanisms of Treatment Outcome in Chronic Pain: Evidence From Routine Care. Front Psychiatry. 2021 Aug 3;12:617871. doi: 10.3389/fpsyt.2021.617871. eCollection 2021. PMID 34413794
- [Background] Dikmen HA, Terzioglu F. Effects of Reflexology and Progressive Muscle Relaxation on Pain, Fatigue, and Quality of Life during Chemotherapy in Gynecologic Cancer Patients. Pain Manag Nurs. 2019 Feb;20(1):47-53. doi: 10.1016/j.pmn.2018.03.001. Epub 2018 Dec 13. PMID 29776873
- [Background] Darnall BD, Carr DB, Schatman ME. Pain Psychology and the Biopsychosocial Model of Pain Treatment: Ethical Imperatives and Social Responsibility. Pain Med. 2017 Aug 1;18(8):1413-1415. doi: 10.1093/pm/pnw166. No abstract available. PMID 27425187
- [Background] Al Hasbi, H., Chayati, N., & Makiyah, S. N. N. (2019). Progressive muscle relaxation to reduces chronic pain in hemodialysis patient. MEDISAINS: Jurnal Ilmiah Ilmu-Ilmu Kesehatan, 17(3), 62-66.
- [Background] Elamin S, E Elbasher AH, E Ali SE, Abu-Aisha H. Arabic translation, adaptation, and validation of the kidney disease quality of life short-form 36. Saudi J Kidney Dis Transpl. 2019 Nov-Dec;30(6):1322-1332. doi: 10.4103/1319-2442.275476. PMID 31929279
- [Background] Alhawatmeh H, Albataineh R, Abuhammad S. Differential effects of guided imagery and progressive muscle relaxation on physical and emotional symptoms in nursing students taking initial clinical training: A randomized clinical trial. Heliyon. 2022 Oct 19;8(10):e11147. doi: 10.1016/j.heliyon.2022.e11147. eCollection 2022 Oct. PMID 36311359